CLINICAL TRIAL: NCT05810220
Title: Investigating Auditory Processing in the Users of Auditory Brainstem and Cochlear Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Cochlear Americas (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-00323
Record Dates: First submitted 2023-03-20; First posted 2023-04-12 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hearing-Impaired Individuals who use Cochlear Implants or Auditory Brainstem Implant (ABI) Devices (Experimental): Two types of measurements will be obtained:
  1. Perceptual: one or more sounds are presented and a behavioral response is collected (e.g., judgements of loudness, pitch or other differences between the sounds, or identifying the word or sentence that was said).
  2. Physiological: noninvasive electrophysiological recordings of nervous system activity.
  Interventions: Device: Electrode-Neural Interface

INTERVENTIONS:
Device: Electrode-Neural Interface — Measurements taken from the electrode-neural interface will be used to guide elimination of poorly functioning ABI electrodes and improve speech perception outcomes.

SUMMARY:
This is a basic investigational research study conducted with hearing impaired adults and children who use cochlear implant or auditory brainstem implant (ABI) devices. The study will evaluate different aspects of hearing and auditory processing in the users of implantable auditory devices.

ELIGIBILITY:
Inclusion Criteria:

* Hearing impaired adult and or child (above 2 years old) who uses ABIs or cochlear implants.
* No diagnosis of any other communicative or cognitive disorder other than hearing impairment. The individual must be able to visit the lab in order to participate in behavioral and electrophysiological experiments.
* Patients' implant device must have useable electrodes that do not result in uncomfortable or unpleasant non-auditory sensation.

Exclusion Criteria:

* Diagnosed cognitive or communicative disorders (other than hearing impairment)
* Severe neurological disorders
* No useable electrodes in their implants

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-12-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percent of Correctly-Identified Speech Materials | Day 1 (Visit 1 - Average visit length is about 3 hours)
  Participants will listen to speech sounds and indicate what sentence or word they heard. The outcome is the percent of speech sounds that are correctly identified.
Percent of Correctly-Identified Stimuli Characteristics when Two or More Stimuli are Presented | Day 1 (Visit 1 - Average visit length is about 3 hours)
  Two or more stimuli will be presented to participants, who will indicate which one is louder, which is higher pitched, or which one is different. The outcome is the percent of stimuli characteristics that are correctly identified.

CONTACTS AND LOCATIONS:
Overall Officials: Mahan Azadpour, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [Mahan.Azadpour@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Mahan.Azadpour@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.